CLINICAL TRIAL: NCT01268163
Title: A Phase 1, Double-blinded, Randomised, Multi-centre, Three-period, Three-treatment, Crossover Study to Compare the Intravenous Pharmacokinetic and Safety Characteristics of European Taxotere® and American Taxotere® With Hospira Docetaxel Injection Administered at a Therapeutic Dose in Cancer Patients.
Brief Title: The Pharmacokinetics and Safety Characteristics of Docetaxel in Patients With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DOE061
Record Dates: First submitted 2010-10-08; First posted 2010-12-29 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2015-07

CONDITIONS: Cancer
Keywords: Docetaxel; Phase I; Pharmacokinetic; Bioequivalence
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): European Taxotere® (Taxotere EU) 60-100 mg/m^2
  Interventions: Drug: European Taxotere®
- 3 (Experimental): Hospira Docetaxel Injection 60-100 mg/m^2
  Interventions: Drug: Hospira Docetaxel Injection
- 2 (Active Comparator): American Taxotere® (Taxotere US) 60-100 mg/m^2
  Interventions: Drug: American Taxotere®

INTERVENTIONS:
Drug: European Taxotere® — 60-100 mg/m^2 IV
  Arms: 1
Drug: American Taxotere® — 60-100 mg/m^2 IV
  Arms: 2
Drug: Hospira Docetaxel Injection — 60-100 mg/m^2 IV
  Arms: 3

SUMMARY:
The purpose of this study is to compare the pharmacokinetic and safety characteristics of European Taxotere® and American Taxotere® with Hospira Docetaxel injection in patients with cancer.

DETAILED DESCRIPTION:
No information is available on the pharmacokinetic characteristics, safety or efficacy of Hospira Docetaxel Injection. The primary purpose of this study therefore is to compare the pharmacokinetic characteristics of 60-100 mg/m² Hospira Docetaxel Injection, 60-100 mg/m² European Taxotere® (Taxotere® EU) and 60-100 mg/m² American Taxotere® (Taxotere® US) when administered as a 1 hour intravenous infusion in man. The secondary objective of this study will be to compare the safety and tolerability of Hospira Docetaxel Injection, Taxotere® EU and Taxotere® US. The study will also provide an opportunity to assess selected efficacy endpoints according to local practice after each cycle of treatment.

The study dosing regimen (60-100 mg/m², administered as a 1 hour intravenous infusion at 3 week intervals) and subject population (cancer patients for whom Taxotere® monotherapy would be a suitable treatment option) were selected on the basis of the licensed use of 60-100 mg/m² Taxotere®. The randomised crossover design was chosen to reduce the effect of intersubject variation.

Since Hospira Docetaxel Injection has not been administered to man there is no information on the risks associated with its clinical use. However the active ingredient of Hospira Docetaxel Injection is the same as that of Taxotere® and it is expected that Hospira Docetaxel Injection will exhibit a similar safety and tolerability profile.

An estimated 24 patients will be recruited at several United Kingdom sites and one Russian site to provide 19 evaluable patients

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent given;
* Have medically documented cancer for which Taxotere® monotherapy would be a suitable treatment option;
* Aged ≥18 years;
* Eastern Cooperative Oncology Group (ECOG) performance status between 0 - 1 (inclusive);
* Haematological and serum chemical parameters that comply with the following criteria (based on local laboratory normal reference range):

  * Haemoglobin ≥9.5 g/dL
  * Leukocytes ≥3.0 x 10^9/L
  * Neutrophils ≥1.5 x 10^9/L
  * Platelets ≥100 x 10^9 L
  * Total bilirubin ≤2.0 x Upper Limit of Normal (ULN)
  * Aspartate aminotransferase (AST) ≤2.5 x ULN
  * Alanine aminotransferase (ALT) ≤2.5 x ULN
  * Alkaline phosphatase ≤4.0 x ULN
  * Serum creatinine ≤1.5 x ULN
* Willing to use an effective method of contraception, i.e. intrauterine device (IUD), oral contraceptive, subdermal implant or double barrier (condom with a contraceptive sponge or contraceptive suppository), unless anatomically sterile, from screening until at least 12 weeks after last dose of Investigational Medicinal Product.
* Willing and able to comply with the requirements of the protocol and available for the planned duration of the study.

Exclusion Criteria:

* Concomitant treatment with any other cytotoxic agent;
* Concomitant use of compounds that induce, inhibit or are metabolized by cytochrome P450, e.g. ciclosporin, ketoconazole, erythromycin, St John's Wort;
* History or presence of any clinically significant findings that, in the opinion of the Investigator, would preclude inclusion in the study;
* Clinically significant vital signs or 12-lead electrocardiogram (ECG) results, as judged by the Investigator;
* Participation in any other clinical trial using an Investigational Medicinal Product within the previous month
* History of Hepatitis B Virus, Hepatitis C Virus or Human Immunodeficiency Virus;
* Recent or clinically significant history of drug or alcohol abuse;
* Insulin-dependent or unstable Diabetes Mellitus;
* History of severe hypersensitivity reactions to Taxotere® or to other drugs formulated with Polysorbate 80;
* History of reaction to any drug containing polyethylene glycol 300 (PEG 300);
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Area under the concentration time curve from zero to last measured concentration (AUC[0-tlast]) | On Day 1, 2, 3, 22, 23, 24, 43, 44, 45 (pre-dose and 30 min, 58 min, 65 min, 70 min, 90 min, 2 hr, 3 hr, 5 hr, 7 hr, 24±2 hr and 48±2 hr after starting Investigational medicinal product infusion during each treatment cycle).
Maximum plasma concentration observed (Cmax) | On Day 1, 2, 3, 22, 23, 24, 43, 44, 45 (pre-dose and 30 min, 58 min, 65 min, 70 min, 90 min, 2 hr, 3 hr, 5 hr, 7 hr, 24±2 hr and 48±2 hr after starting Investigational medicinal product infusion during each treatment cycle).

SECONDARY OUTCOMES:
Area under the concentration time curve from zero to infinity (AUC0-∞) | On Day 1, 2, 3, 22, 23, 24, 43, 44, 45 (pre-dose and 30 min, 58 min, 65 min, 70 min, 90 min, 2 hr, 3 hr, 5 hr, 7 hr, 24±2 hr and 48±2 hr after starting Investigational medicinal product infusion during each treatment cycle).
Terminal elimination half life (t1/2) | On Day 1, 2, 3, 22, 23, 24, 43, 44, 45 (pre-dose and 30 min, 58 min, 65 min, 70 min, 90 min, 2 hr, 3 hr, 5 hr, 7 hr, 24±2 hr and 48±2 hr after starting Investigational medicinal product infusion during each treatment cycle).
Elimination rate constant (Kel) | On Day 1, 2, 3, 22, 23, 24, 43, 44, 45 (pre-dose and 30 min, 58 min, 65 min, 70 min, 90 min, 2 hr, 3 hr, 5 hr, 7 hr, 24±2 hr and 48±2 hr after starting Investigational medicinal product infusion during each treatment cycle).
Total plasma clearance (CL) | On Day 1, 2, 3, 22, 23, 24, 43, 44, 45 (pre-dose and 30 min, 58 min, 65 min, 70 min, 90 min, 2 hr, 3 hr, 5 hr, 7 hr, 24±2 hr and 48±2 hr after starting Investigational medicinal product infusion during each treatment cycle).
Volume of distribution (Vss) | On Day 1, 2, 3, 22, 23, 24, 43, 44, 45 (pre-dose and 30 min, 58 min, 65 min, 70 min, 90 min, 2 hr, 3 hr, 5 hr, 7 hr, 24±2 hr and 48±2 hr after starting Investigational medicinal product infusion during each treatment cycle).
Area under the concentration time curve for unbound docetaxel | On Day 1, 2, 3, 22, 23, 24, 43, 44, 45 (pre-dose and 30 min, 58 min, 65 min, 70 min, 90 min, 2 hr, 3 hr, 5 hr, 7 hr, 24±2 hr and 48±2 hr after starting Investigational medicinal product infusion during each treatment cycle).

CONTACTS AND LOCATIONS:
Overall Officials: M. Ranson, Principal Investigator — Christie Hospital, Manchester; V Semiglazov, Principal Investigator — N.N. Petrov Research Institute of Oncology
Locations (4):
- Saint Petersburg, Russia
- United Kingdom (3):
  - Cambridge
  - Glasgow
  - Manchester